CLINICAL TRIAL: NCT01326754
Title: Efficacy and Safety of the Dispersible Formulation of Artemether-lumefantrine, Co-formulated Artesunate-amodiaquine and Co-formulated Dihydroartemisinin-piperaquine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Machinga District, Malawi
Brief Title: Efficacy of Artemether-lumefantrine, Artesunate-amodiaquine and Dihydroartemisinin-piperaquine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jacek Skarbinski, Medical Epidemiologist, Centers for Disease Control and Prevention
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-CGH-6029
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artemether-lumefantrine (Other)
  Interventions: Drug: Artemether-lumefantrine combination
- Artesunate-amodiaquine (Other)
  Interventions: Drug: Artesunate-amodiaquine combination
- Dihydroartemisinin-piperaquine (Other)
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — Dispersible formulation of artemether-lumefantrine at a dose of 2/12 mg/kg body weight of artemether and lumefantrine, respectively, per dose, given twice a day for 3 days
  Arms: Artemether-lumefantrine
Drug: Artesunate-amodiaquine combination — Co-formulated artesunate-amodiaquine at a dose of 4 mg/kg/day artesunate and 10 mg/kg/day amodiaquine once a day for 3 days
  Arms: Artesunate-amodiaquine
Drug: Dihydroartemisinin-piperaquine — Co-formulated dihydroartemisinin-piperaquine at a dose of 4 mg/kg/day dihydroartemisinin and 18 mg/kg/day piperaquine once a day for 3 days
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Background: Malaria is a cause of substantial morbidity and mortality in Malawi. Prompt and effective treatment of uncomplicated malaria remains a key strategy to reduce the public health burden of malaria. Due to the rising resistance to and falling efficacy of sulfadoxine-pyrimethamine, the first-line treatment of uncomplicated malaria from 1993 to 2007, the National Malaria Control Program (NMCP) revised the national treatment guidelines in 2007. The revised treatment guidelines recommend artemether-lumefantrine as the first-line treatment for uncomplicated malaria and artesunate-amodiaquine as a second-line treatment for uncomplicated malaria. The change in policy was based primarily on efficacy data from other countries in sub-Saharan Africa. However, although both artemether-lumefantrine and artesunate-amodiaquine have been in use in Malawi since 2007, there are relatively few studies assessing their efficacy. In a study conducted in 2004-2006 in Blantyre, artemether-lumefantrine was found to be efficacious.1 In addition, a more recent assessment of artemether-lumefantrine in vivo efficacy conducted in six sites in Malawi in 2009 also suggests that the standard formulation artemether-lumefantrine remains highly efficacious (Kamija Phiri, personal communication).

Although, some Malawi-specific data on the in vivo efficacy of the standard formulation of artemether-lumefantrine exists, there are additional data that is needed to support the current policy and inform future policy decisions. In 2010 the NMCP has introduced the dispersible formulation of artemether-lumefantrine (Coartem-D™) for use as a first-line antimalarial in Malawi, due to the global unavailability of the standard formulation of artemether-lumefantrine from Novartis, the key supplier of the standard formulation of artemether-lumefantrine (Coartem™) in Malawi. In light of these developments, an assessment of the efficacy, safety and tolerability of the dispersible formulation of artemether-lumefantrine is warranted. In addition, the efficacy, safety and tolerability of co-formulated artesunate-amodiaquine, the current secondline treatment for uncomplicated malaria, has never been assessed in Malawi and should be evaluated. Lastly, dihydroartemisinin-piperaquine has recently been added to the new World Health Organization (WHO) guidelines for the treatment of uncomplicated malaria. This promising new antimalarial might have a role as a first-line or second-line antimalarial for the treatment of uncomplicated malaria, but there are no efficacy and safety data from Malawi. This knowledge gap needs to be addressed to help inform policy makers about the potential role of dihydroartemisinin-piperaquine for the treatment of uncomplicated malaria in Malawi.

Objective: Efficacy and safety of the dispersible formulation of artemether-lumefantrine, co-formulated artesunate-amodiaquine and co-formulated dihydroartemisinin-piperaquine for the treatment of uncomplicated Plasmodium falciparum malaria at Machinga District Hospital- Malawi

Methods: An antimalarial drug efficacy trial will be conducted in Malawi. The participants will be febrile people 6-59 months old with confirmed uncomplicated P. falciparum infection. Patients will be sequentially allocated to receive treatment with either the dispersible formulation of artemether-lumefantrine at a dose of 2/12 mg/kg body weight of artemether and lumefantrine, respectively, per dose, given twice a day for 3 days; or co-formulated artesunate-amodiaquine at a dose of 4 mg/kg/day artesunate and 10 mg/kg/day amodiaquine once a day for 3 days; or co-formulated dihydroartemisinin-piperaquine at a dose of 4 mg/kg/day dihydroartemisinin and 18 mg/kg/day piperaquine once a day for 3 days. Clinical and parasitological parameters will be monitored over a 42-day follow-up period to evaluate drug effi¬cacy. The study will be conducted from January to December, 2011. The results of this study will be used to assist the Ministry of Health in Malawi in assessing the current national treatment guidelines for uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 to 59 months;
* mono-infection with P. falciparum detected by microscopy;
* parasitaemia of 2,000-200,000/µl asexual forms;
* presence of axillary or tympanic temperature ≥ 37.5 °C or oral or rectal temperature of ≥ 38 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* informed consent from the parent or guardian of the child.

Exclusion Criteria:

* presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO (Appendix 1);
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition (defined as a child whose growth stand¬ard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm) and calculated using EpiInfo 2002 EpiNut calculator;
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s).

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 498 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response (ACPR) | 42 days
  Absence of parasitaemia on day 42, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Skarbinski, MD, Principal Investigator — Centers for Disease Control and Prevention; Don Mathanga, MBBS PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Machinga District Hospital, Liwonde, Malawi